CLINICAL TRIAL: NCT00003719
Title: Phase II Evaluation of Irinotecan (CPT-11) in Previously Treated Advanced Sarcomas
Brief Title: Irinotecan in Treating Patients With Stage IV or Recurrent Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066828; CPMC-IRB-8100; NCI-V98-1511
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2001-08

CONDITIONS: Sarcoma
Keywords: stage IV adult soft tissue sarcoma; recurrent adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Irinotecan

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irinotecan in treating patients who have stage IV or recurrent soft tissue sarcoma that has been previously treated with chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of irinotecan in patients with metastatic, recurrent, or unresectable locally advanced previously treated soft tissue sarcoma. II. Assess the clinical and laboratory toxic effects and patient tolerance of this regimen in these patients.

OUTLINE: Patients receive irinotecan IV over 90 minutes weekly for 4 weeks, followed by 2 weeks of rest. Treatment continues every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for the first two years, then every 6 months for the next two years, and every 12 months thereafter until death.

PROJECTED ACCRUAL: A total of 14-27 patients will be accrued for this study in 18-36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed recurrent or stage IV (metastatic or locally advanced) unresectable soft tissue sarcoma Patients with soft tissue Ewing's sarcoma, Kaposi's sarcoma, sarcoma of the bone, and mesothelioma are not eligible Must have failed at least one, but no more than two, prior chemotherapy regimens, one of which contained doxorubicin either as adjuvant therapy or first-line therapy for metastatic disease Bidimensionally measurable disease on x-ray, MRI or CT scan, or physical exam (outside of previously irradiated area) No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: Platelet count at least lower limit of normal WBC at least 3,500/mm3 OR Absolute neutrophil count at least 1,750/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL AST no greater than 3 times upper limit of normal (ULN) (no greater than 5 times ULN with liver tumor involvement) Renal: Creatinine less than ULN OR Creatinine clearance greater than 60 mL/min Calcium less than ULN Cardiovascular: No myocardial infarction within past 6 months No congestive heart failure requiring therapy Other: Not pregnant or nursing Fertile patients must use effective contraception No physical, mental, or emotional disorders No other prior malignancy within the past 5 years, except: Adequately treated basal or squamous cell skin cancer Carcinoma in situ of the cervix Adequately treated stage I or II cancer in complete remission No active or uncontrolled infection HIV negative No known Gilbert's syndrome No uncontrolled diabetes (random blood sugar at least 200 mg)

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior biologic response modifier therapy allowed Chemotherapy: See Disease Characteristics No prior irinotecan or topotecan No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy Radiotherapy: See Disease Characteristics At least 3 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: At least 4 weeks since prior surgery and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 1997-07

CONTACTS AND LOCATIONS:
Overall Officials: Robert N. Taub, MD, PhD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center, New York, New York, United States